CLINICAL TRIAL: NCT02136394
Title: Investigation Into the Role of Gastroesophageal Reflux in Pulmonary Fibrosis in Scleroderma
Brief Title: The Role of Gastroesophageal Reflux in Scleroderma Pulmonary Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2013OE006B
Record Dates: First submitted 2013-12-30; First posted 2014-05-13 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Interstitial Lung Disease; Systemic Sclerosis; Gastroesophageal Reflux
MeSH Terms: conditions — Lung Diseases, Interstitial; Scleroderma, Systemic; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Severe/moderate acid reflux
  Interventions: Other: Gastro-esophageal reflux
- Mild/absent acid reflux

INTERVENTIONS:
Other: Gastro-esophageal reflux — This is an observational study. The exposure is the gastro-esophageal reflux.
  Groups: Severe/moderate acid reflux

SUMMARY:
Scarring of the lungs is common in patients with scleroderma and is one of the main causes of death. Patients with scleroderma very frequently have problems with their gullet (esophagus), the food pipe that leads into the stomach.

Normally, a small circular muscle at the base of the esophagus opens to allow food to pass into the stomach and closes to keep the digestive fluids from flowing back up into the gullet. In patients with scleroderma, the muscle may become weak and no longer close properly. Gastroesophageal reflux (GER) is the medical term for reflux of stomach contents into the esophagus.

Our hypothesis is that small amounts of GER can move back up into the esophagus and get inhaled into the lungs, and may be one of the triggers for lung scarring. We propose to look for certain substances normally only found in the stomach in the "exhaled breath condensate" which is collected by breathing comfortably into a cooled cylinder, allowing the breath to condensate. In a smaller group of patients, we also plan to perform a bronchoalveolar lavage, a more widely studied test in which a small amount of fluid is introduced into a small part of the lungs through a fine tube, and then removed for examination, to evaluate whether the two tests provide similar measurements. We will also evaluate the correlation between these molecules and other tests, including lung function, and markers of lung scarring activity, and tests to look at how the esophagus is working so that we can get a clearer picture of how this affects patients' daily lives. Finally, we will be following up patients over time with lung function to see whether evidence of GER into the lungs is linked with a greater likelihood of worsening of lung scarring in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 years
* Diagnosis of SSc (American College of Rheumatology criteria)
* Interstitial lung disease (>5% extent of ILD on HRCT)
* Only for bronchoscopy: presence of troublesome cough and/or GER symptoms and/or recurrent chest infections and/or asymmetry of ILD changes on CT

Exclusion Criteria:

* Significant communication difficulties
* Unable to perform reliable lung function tests
* Current smokers
* Only for bronchoscopy: FEV1 less than 1L or DLCO less than 30% of the predicted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen in the department of respiratory medicine or rheumatology of two teaching hospitals in London.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-12 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Measurements of pepsin and pH in the Exhaled breath condensate (EBC) | Baseline
In a subgroup pf 40 patients, measurements of pepsin and bile salts in bronchoalveolar lavage (BAL) | Baseline
Serum KL-6 | Baseline
  Serum KL-6 is a known marker of alveolar epithelial damage in SSc-ILD
Measurements of pepsin and pH in the Exhaled breath condensate (EBC) | 12 months

SECONDARY OUTCOMES:
Changes from baseline in longitudinal lung function assessment | Baseline, month 6, month 12, month 18
  Spirometry with total lung capacity, diffusing capacity for CO

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Royal free hospital, London
  - Royal Brompton hospital, London